CLINICAL TRIAL: NCT03122327
Title: Comprehensive Geriatric Assessment (cGA) in Newly-diagnosed Elderly Multiple Myeloma (MM) Patients: a Multi-center, Prospective, Non-interventional Study.
Brief Title: cGA in Newly-diagnosed Elderly MM Patients: a Multi-center, Prospective, Non-interventional Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jian Li, Associated professor in hematology, Peking Union Medical College Hospital
Other Study IDs: S-K230
Record Dates: First submitted 2017-04-18; First posted 2017-04-20 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma; Comprehensive Geriatric Assessment
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly diagnosed MM patients: newly diagnosed MM patients who fulfilled the inclusion criteria for this study
  Interventions: Other: Questionaires

INTERVENTIONS:
Other: Questionaires — Questionaires of cGA assessment. No other interventions would be carried out aside from the standard treatment for MM.

SUMMARY:
This is a multi-center, prospective, non-interventional study. Eligible newly diagnosed elderly multiple myeloma (MM) patients will receive comprehensive geriatric assessment (cGA) including ECOG scale, questionaires of ADL（activities of daily living), IADL(instrumental ADL),MNA-SF(mini-nutritional assessment), GDS(geriatric depression scale), MMSE(mini-mental state examination), SF-36 and CCI (charlson comorbidity index). Patients will get standard care for MM and receive the above assessments at baseline and after cycle 1, 4 and 12 for treating MM.Follow-up information and survival data of these MM patients would be collected. We would evaluate the cGA status of these newly diagnosed elderly MM patients and investigate the association of cGA parameters with patient's survival.

DETAILED DESCRIPTION:
Baseline: ECOG, ADL, IADL, MNA-SF, GDS, MMSE, SF-36 and CCI; After cycle 1: ECOG,ADL,IADL,GDS and SF-36 After cycle 4: ECOG,ADL,IADL,GDS, MNA-SF and SF-36 After cycle 12: ECOG,ADL,IADL,GDS, MNA-SF and SF-36

ELIGIBILITY:
Inclusion Criteria:

* age>=65 years old;
* newly diagnosed and untreated MM patients;
* able to provide informed consent

Exclusion Criteria:

* refused to participate;
* with concomitant amyloidosis;
* smoldering MM.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Newly diagnosed Multiple myeloma (MM) patients>=65 years old
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Current status of cGA in newly diagnosed elderly MM patients | 12 cycles of MM treatment (about 12 months) after the last patient begins treatment
  Description of the cGA (comprehensive geriatric assessment) status of the target population which is currently not known in China. The cGA parameters to be described include baseline ECOG, ADL（activities of daily living), IADL(instrumental ADL),MNA-SF(mini-nutritional assessment), GDS(geriatric depression scale), MMSE(mini-mental state examination), SF-36 and CCI (charlson comorbidity index) which would be carried out by trained physicians. The physicians would receive standard training from geriatricians of Peking Union Medical College Hospital. Moreover, as the treatment for MM (multiple myeloma) patients continues, re-evaluation of the cGA parameters would be done. The status of ECOG, ADL, IADL, GDS, SF-36 would be re-evaluated after cycle 1, 4, 12 of MM treatment. And MNA-SF scale would be re-assessed after cycle 4 and 12 of MM treatment. A description of the changes of the above scales would also be recorded for these MM patients.

SECONDARY OUTCOMES:
Association between the baseline cGA parameters and patients' overall survival | 5 years after the last patient begins treatment for MM
  To evaluate the association of the baseline cGA parameters (including ECOG, ADL, IADL,MNA-SF, GDS, MMSE, SF-36 and CCI ) and patient's overall survival
Association between baseline cGA parameters and patients' progression free survival | 5 years after the last patient begins treatment for MM
  To evaluate the association of cGA parameters (including ECOG, ADL, IADL,MNA-SF, GDS, MMSE, SF-36 and CCI ) and patient's progression free survival

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Derived] Yao Y, Sui WW, Liao AJ, Wang W, Chen LJ, Chu XX, Bao L, Cen XN, Fu R, Liu H, Sun CY, Jin FY, Yan H, Wang LQ, Yuan CL, Gao GX, Gao D, Zhang JQ, He JX, Hu JD, Ma LM, Zhang L, Zhou DB, Zou DH, Li J. Comprehensive geriatric assessment in newly diagnosed older myeloma patients: a multicentre, prospective, non-interventional study. Age Ageing. 2022 Jan 6;51(1):afab211. doi: 10.1093/ageing/afab211. PMID 34673897